CLINICAL TRIAL: NCT02468960
Title: Optimal Lesion Preparation With Non-compliant Balloons for the Implantation of Bioresorbable Vascular Scaffolds (BVS) -OPRENBIS Study
Brief Title: Optimal Lesion Preparation With Non-compliant Balloons Before Implantation Of Bioresorbable Scaffolds (OPreNBiS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SIS Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPreNBiS
Record Dates: First submitted 2015-03-04; First posted 2015-06-11 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Angina; Unstable Angina; Stable Angina
Keywords: Coronary Artery Disease; OPN NC; Angina; Stable; Unstable
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Angina, Unstable; Angina, Stable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPN strategy (study group) (Other): Interventions planned in this arm are as follows:
  * Predilatation with OPN NC balloon catheter.
  * Absorb BVS implantation.
  * Treated segment visualization by OCT.
  * Clinical FU at 12 months.
  Interventions: Device: Predilatation with OPN NC balloon catheter.; Device: Absorb BVS implantation.; Procedure: Treated segment visualization by OCT.; Other: Clinical FU at 12 months.
- Standard strategy (control group) (Other): Interventions planned in this arm are as follows:
  * Predilatation with standard compliant balloon.
  * Absorb BVS implantation.
  * Treated segment visualization by OCT.
  * Clinical FU at 12 months.
  Interventions: Device: Predilatation with standard compliant balloon.; Device: Absorb BVS implantation.; Procedure: Treated segment visualization by OCT.; Other: Clinical FU at 12 months.

INTERVENTIONS:
Device: Predilatation with OPN NC balloon catheter. — Target lesion will be prepared by predilatation with OPN NC balloon catheter.
  Arms: OPN strategy (study group)
Device: Predilatation with standard compliant balloon. — Target lesion will be prepared by predilatation with standard balloon catheter (compliant).
  Arms: Standard strategy (control group)
Device: Absorb BVS implantation. — After lesion preparation implantation of BVS Absorb scaffold will be performed.
Procedure: Treated segment visualization by OCT. — Finally treated segment will be visualized by Intravascular Optical Coherence Tomography (OCT).
Other: Clinical FU at 12 months. — All patients will be clinically followed for 12 months.

SUMMARY:
Study aim : To compare a novel strategy of lesion preparation with noncompliant balloons before implantation of BVS (Bioresorbable Vascular Scaffold).

Hypothesis: Predilatation with non-compliant balloons could facilitate optimal deployment of BVS. By achieving good scaffold apposition a need for post-dilatation could be significantly reduced. This is expected to result in better short- and long-term outcomes.

DETAILED DESCRIPTION:
Study design:

Following pre-dilatation a BVS will be implanted and optical coherence tomography (OCT) will be performed in all patients. After OCT post-dilatation with non-compliant balloons might be performed if this is considered necessary by the treating interventionist. Final OCT will be performed in all patients. 1:1 Randomization of two strategies before the implantation of bioresorbable scaffolds:

* OPN strategy (study group): pre-dilatation with OPN NC ® Super High Pressure PTCA (Percutaneous Transluminal Coronary Angioplasty) balloons
* standard strategy (control group): pre-dilatation with a standard (compliant) balloon

Enrolment:

Randomization of 50 patients

* 25 in the OPN strategy (study group)
* 25 in the standard strategy (control group)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Able and willing to give informed consent.
* Willing to comply with specified follow-up evaluations.
* Clinical manifestation of coronary artery disease: stable angina, unstable angina or non-ST-elevation myocardial infarction.
* De novo lesion.
* Angiographic diameter stenosis > 70 % and/or fractional flow reserve <0.80.
* Vessel diameter between 2.5 and 4.0 mm.
* One- or two vessel disease (defined as diameter stenosis > 70 % in vessels with a diameter > 2.5 mm).
* Up to two lesions in one or two vessels can be treated

Exclusion Criteria:

* Patient characteristics

  * Pregnant or nursing patient or planned pregnancy in the period up to 1 year following the index procedure.
  * Patient with contraindication for 12 months of dual antiplatelet therapy.
  * ST-elevation myocardial infarction.
  * Any contraindication to the implantation of BVS. Lesion characteristics
  * Visible thrombus in coronary angiography
  * Chronic total occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Scaffold apposition ratio in both groups (ratio of malapossition stents to total stents per cross-section | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
  Outcome will be analyzed by independent Angio CoreLab based on data recorded during index PCI procedure.

SECONDARY OUTCOMES:
Procedural success defined as successful delivery of the scaffold | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Need for post-dilatation after implantation of the scaffold | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
Scaffold apposition after post-dilatation | Participants will be followed for the duration of index procedure, an expected average of 1 hour.
  Outcome will be analyzed by independent Angio CoreLab based on data recorded during index PCI procedure.
Frequency and total number of periprocedural complications: dissection, slow- or no flow, dissection requiring additional stent implantation, | Participants will be followed for the duration of index procedure, an expected average of 1 hour.

OTHER OUTCOMES:
Number of patients with diagnosis of periprocedural myocardial infarction defined as 5x upper reference level elevation of high sensitive Troponin I (in patients with normal pre-procedural Troponin) | Participants will be followed for the duration of hospital stay, an expected average of 5 days.
Number of patients with diagnosis of in-stent restenosis requiring revascularization within 12 months post-procedure | 12 month folow up
Rate of stent thrombosis according the ARC criteria within 12 months post procedure | 12 month follow up
Death or myocardial infarction within 12 months post-procedure | 12 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, Prof. dr, Principal Investigator
Locations (1):
- Luzernen Kantonsspital, Spitalstrasse 16, Lucerne, Switzerland